CLINICAL TRIAL: NCT04919408
Title: Evaluation of the Incidence of Chronic Post-cesarean Pain as Part of an Enhanced Recovery After Surgery (ERAS) Protocol.
Acronym: ChroCéRAAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021-CHITS-003; 2021-A00397-34 (Other: IdRCB)
Record Dates: First submitted 2021-06-01; First posted 2021-06-09 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Chronic Post-cesarean Pain
Keywords: Chronic pain; Enhanced Rehabilitation After Surgery; Cesarean section; Persistant pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients scheduled for cesarean section under spinal anesthesia (Experimental): Patients scheduled for cesarean section under spinal anesthesia ASA I and II according to The ASA Physical Status Classification System
  Interventions: Other: telephone survey

INTERVENTIONS:
Other: telephone survey — telephone survey with a questionnaire to assess pain at 3 months and then 6 months after their cesarean section

SUMMARY:
Enhanced Rehabilitation After Surgery (ERAS), developed in the 1990s, is a program encompassing a set of measures before, during and after surgery aimed at improving management by promoting the early recovery of the patient's abilities after surgery.

The ERAS has been scientifically validated and standardized in many surgical disciplines since the implementation of guidelines in France in 2016.

Regarding the obstetrical field, it was not until 2018 that the caesarean section could benefit from ERAS, with the publication of specific guidelines.

Several studies have been able to demonstrate ERAS effectiveness in reducing the length of hospitalization, postoperative complications, the consumption of analgesics immediately after surgery, and the financial cost, including in the context of cesarean sections.

But beyond immediate benefit, the impact of an ERAS protocol on chronic pain has not yet been evaluated.

Chronic pain is defined as physical discomfort that persists for more than 2 months after surgery.

It was not until 2004 that research focused on chronic post-cesarean pain, finding an incidence of chronic pain of 18.6% at 3 months and 12.3% at 6 months. In 2016, another study estimated an incidence of chronic pain in the caesarean scar at 15% at 3 months and 11% at 1 year. The investigators can notice that the presence of chronic post-cesarean pain remained stable over this period.

Several risk factors have been identified, such as the presence of acute pain immediately after surgery, the type of anesthesia, the type of surgical incision or a significant state of anxiety before the operation.

In this context, the investigators wish to assess the rate of chronic post-surgical pain in scheduled cesarean sections (excluding emergencies) under spinal anesthesia as part of a ERAS protocol. The investigatrors will also specify the type of pain and its impact on the daily activities of young mothers and will assess the level of adherence of medical and paramedical teams to the ERAS protocol.

To answer these questions, the investigators will conduct a telephone survey with a questionnaire to assess pain at 3 months and then 6 months after their cesarean section. The pain studied is defined as being the pain at the level of the caesarean scar.

This is an innovative subject evaluating the impact of the implementation of an ERAS protocol on chronic pain. Depending on the results, the investigators will be able to optimize the prevention of chronic pain of cesarean section.

DETAILED DESCRIPTION:
Enhanced Rehabilitation After Surgery (ERAS), developed in the 1990s, is a program encompassing a set of measures before, during and after surgery aimed at improving management by promoting the early recovery of the patient's abilities after surgery.

The ERAS has been scientifically validated and is currently standardized in many surgical disciplines since the implementation of guidelines in France in 2016.

Regarding the obstetrical field, it was not until 2018 that the caesarean section could benefit from ERAS, with the publication of specific guidelines.

Several studies have been able to demonstrate ERAS effectiveness in reducing the length of hospitalization, postoperative complications, the consumption of analgesics immediately after surgery, and the financial cost, including in the context of cesarean sections.

But beyond immediate benefit, the impact of an ERAS protocol on chronic pain has not yet been evaluated.

Chronic pain is defined as physical discomfort that persists for more than 2 months after surgery.

It was not until 2004 that research focused on chronic post-cesarean pain, finding an incidence of chronic pain of 18.6% at 3 months and 12.3% at 6 months. In 2016, another study estimated an incidence of chronic pain in the caesarean scar at 15% at 3 months and 11% at 1 year. The investigators can notice that the presence of chronic post-cesarean pain remained stable over this period.

Several risk factors have been identified, such as the presence of acute pain immediately after surgery, the type of anesthesia, the type of surgical incision or a significant state of anxiety before the operation.

In this context, the investigators wish to assess the rate of chronic post-surgical pain in scheduled cesarean sections (excluding emergencies) under spinal anesthesia as part of a ERAS protocol. The investigatrors will also specify the type of pain and its impact on the daily activities of young mothers and will assess the level of adherence of medical and paramedical teams to the ERAS protocol.

To answer these questions, the investigators will conduct a telephone survey with a questionnaire to assess pain at 3 months and then 6 months after their cesarean section. The pain studied is defined as being the pain at the level of the caesarean scar.

This is an innovative subject evaluating the impact of the implementation of an ERAS protocol on chronic pain. Depending on the results, the investigators will be able to optimize the prevention of chronic pain of cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for cesarean section under spinal anesthesia
* Patients ASA I and II according to The ASA Physical Status Classification System

Exclusion Criteria:

intervention under general anesthesia

* complication during the operation
* post-partum haemorrrhage
* pre-op anemia <9g / dl
* Patient under judicial protection (guardianship, curatorship...) or safeguard of justice.
* Patient unable to answer the questionnaires by telephone (not speaking French, hard of hearing, mute French language, hearing impaired, mute...)
* Any other reason that, in the opinion of the investigator, could interfere with the evaluation of the objectives of the study

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 283 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2024-04-17 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
To study the incidence of chronic post-surgical pain in scheduled cesarean section under spinal anesthesia as part of a ERAS protocol. | 3 months
  The importance of the pain will be assessed using a verbal scale made up of the items : absent, minimal, moderate and severe.
  The incidence rate at 3 months will be calculated as follows:
  Number of patients with minimal, moderate or severe scar pain 3 months after their cesarean section / Number of patients evaluable at 3 months

SECONDARY OUTCOMES:
To study the incidence of chronic post-surgical pain in scheduled cesarean section under spinal anesthesia as part of a ERAS protocol. | 6 months
  The importance of the pain will be assessed using a verbal scale made up of the items : absent, minimal, moderate and severe.
  The incidence rate at 6 months will be calculated as follows:
  Number of patients with minimal, moderate or severe scar pain 6 months after their cesarean section / Number of patients evaluable at 6 months
Specify the type and extent of the pain | 6 months
  The type and extent of the pain will be assessed using a verbal scale adapted from the questionnaire used in the study by L. Nikolajsen et al(1), and the DN4 questionnaire to search for neuropathic pain.
Evaluate the chronical pain impact on daily activities of young mothers | 6 months
  The chronical pain impact on daily activities of young mothers will be assessed using a verbal scale adapted from the questionnaire used in the study by L. Nikolajsen et al(1)
Evaluate the rate of adherence to the ERAS protocol. | 24 months
  As the anesthesiology department is affiliated with the French ERAS society : GRACE (French-speaking group for improved rehabilitation after surgery), we will use their audit tool to assess the rate of adherence to ERAS protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Géraldine SLEHOFER-LHERIAU, MD, Study Director — Anesthesiology department Hôpital Sainte Musse
Locations (2):
- France (2):
  - Hôpital Nord, Marseille, Bouches-du-Rhône
  - Centre Hospitalier Intercommunal Toulon La Seyne sur Mer, Toulon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nikolajsen L, Sorensen HC, Jensen TS, Kehlet H. Chronic pain following Caesarean section. Acta Anaesthesiol Scand. 2004 Jan;48(1):111-6. doi: 10.1111/j.1399-6576.2004.00271.x. PMID 14674981
- See also: As the anesthesia service is affiliated with the French ERAS Society GRACE (French-speaking group for improved rehabilitation after surgery), we will use their audit tool to assess the rate of adherence to ERAS protocol for cesarean section. — https://www.grace-audit.fr/accueil/index.php